CLINICAL TRIAL: NCT07170631
Title: Effectiveness of a General Therapeutic Exercise Program Including Specific Upper Limb Exercises to Reduce Lymphedema and Peripheral Neuropathy Secondary to Oncological Treatment in Patients With Breast Cancer: A Pre-post Intervention Study (LYNMA)
Brief Title: Effectiveness of a Therapeutic Exercise Program With Specific Upper Limb Exercises to Reduce Lymphedema and Neuropathy in Breast Cancer Patients: A Pre-post Study (LYNMA)
Acronym: LYNMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Aïda Cadellans-Arróniz, PhD, Associate Professor, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIS-2025-07
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Lymphedema Arm; Lymphedema Due to Radiation; Lymphedema, Breast Cancer; Peripheral Neuropathy Due to Chemotherapy; Peripheral Neuropathy in Breast Cancer Patient
Keywords: Therapeutic exercise; Breast cancer; Lymphedema; Peripheral neuropathy; Upper limb exercises; Oncology physiotherapy; Neural mobilization; Neurodynamic techniques; Peripheral nerve ultrasound
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms; Lymphedema; Peripheral Nervous System Diseases | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic exercise (Experimental): Participants will undergo a general therapeutic exercise program including specific upper limb exercises designed to reduce lymphedema and neuropathy secondary to cancer treatment. The program consists of supervised sessions two times per week over 12 weeks, led by a specialized physiotherapist. Exercises include mobility, strength, and neurodynamic techniques.
  Interventions: Other: Therapeutic exercise

INTERVENTIONS:
Other: Therapeutic exercise — Participants will follow a 3-month therapeutic exercise program combining general exercises with specific upper limb exercises, including hand proprioception and neurodynamic techniques. Two group sessions per week (1 to 1.15 hours each) will be conducted, with at least 24 hours between sessions. Each session includes warm-up, three progressive work blocks with strength, mobility, and balance exercises, and a cool-down. Strength training uses body weight and equipment, with intensity guided by the Rate of Perceived Exertion (RPE) scale, progressing safely from moderate to higher levels. Mobility and balance exercises target trunk, upper and lower limbs, and postural control. Neurodynamic techniques focus on median, radial, and ulnar nerves using neural sliding and intermittent tension, stopping exercises if pain exceeds 4/10. Supervised by experienced physiotherapists, the program aims to reduce lymphedema and neuropathy symptoms in breast cancer patients undergoing cancer treatment.

SUMMARY:
This study aims to evaluate the effectiveness of a therapeutic exercise program designed specifically for women with breast cancer. The program includes general exercises along with specific movements for the upper limb to help reduce common side effects of cancer treatment such as lymphedema (swelling of the arm) and neuropathy (nerve pain or numbness). Participants will undergo the exercise program and be assessed before and after to determine improvements in their symptoms and overall quality of life. The goal is to provide evidence that targeted physical therapy can improve recovery and well-being in breast cancer survivors.

DETAILED DESCRIPTION:
This pre-post intervention study aims to assess the effectiveness of a comprehensive therapeutic exercise program tailored for breast cancer patients experiencing lymphedema and neuropathy secondary to cancer treatment. The program combines general physical exercises with specific upper limb movements targeting symptom reduction and functional improvement. Participants will be evaluated before and after the intervention to measure changes in arm swelling, nerve symptoms, physical function, and quality of life. The study will contribute valuable data on non-pharmacological rehabilitation strategies that could enhance recovery and reduce long-term complications in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving treatment for breast carcinoma.reatments include surgical procedures (breast-conserving surgery or mastectomy), axillary lymph node dissection, sentinel lymph node biopsy, radiotherapy, chemotherapy, and hormone therapy.
* Participants must provide authorization from their primary care physician and/or oncologist to perform therapeutic exercise.
* Diagnosis of lymphedema associated with stage I or II breast cancer (Stage 1 or mild: circumference difference less than 4 cm [volume difference 10-25%] compared to the healthy arm; Stage 2 or moderate: circumference difference between 4 and 6 cm [volume difference 25-50%] compared to the healthy arm).
* A score of 4 or higher on the DN4 questionnaire (neuropathic pain)

Exclusion Criteria:

* Lack of medical authorization.
* Pre-existing cardiac pathology prior to cancer diagnosis.
* Exacerbation of comorbidities.
* Travel time exceeding 45 minutes to the location where the therapeutic exercise program is conducted.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Excess limb volume (%) compared to the unaffected limb | Baseline (before intervention), Immediately post-program (Day 0 after completion)
  Excess volume of the affected limb (percentage compared to the unaffected limb). The volume of each limb will be measured manually using a measuring tape by taking circumferences every 4 centimeters from the wrist to the axilla. Limb volume will be calculated using the Kuhnke formula: Volume equals the sum of the squares of the circumferences (C1 squared plus C2 squared plus ... plus Cn squared) divided by pi, where C1, C2, … Cn are the circumferences measured at different points along the limb.

SECONDARY OUTCOMES:
Change in neuropathic pain intensity measured with DN4 questionnaire | Baseline (before intervention), Immediately post-program (Day 0 after completion)
  Will be assessed using the DN4 questionnaire, designed to help identify neuropathic pain. It is a simple, quick, and highly reliable tool widely used in clinical practice and research. The questionnaire consists of 10 items divided into two parts: a patient interview and a physical examination performed by the healthcare professional. Each item is scored as "yes" or "no," with each positive answer receiving 1 point. A total score of 4 or more is interpreted as indicative of neuropathic pain
Change in hand grip strength from baseline measured with handheld dynamometer (kg) | Baseline (before intervention), Immediately post-program (Day 0 after completion)
  Hand grip strength will be assessed using a digital hand dynamometer (BIMS). This test is an indicator of overall muscle strength and has been previously used as a marker of clinical and nutritional status, as well as a predictor of decreased functional capacity in breast cancer patients
Change in nerve cross-sectional area measured with high-resolution ultrasound (mm²) | Baseline (before intervention), Immediately post-program (Day 0 after completion)
  Will be assessed using musculoskeletal ultrasound, a useful technique to evaluate possible signs of inflammation, entrapment, or neuropathy. Observed changes can provide relevant information about the presence of inflammation or compression. One common indicator is an increased cross-sectional area of the nerve (measured in mm), which may indicate intraneural edema or an inflammatory process. We will complement the assessment by comparing the affected nerve with the contralateral healthy side to detect differences that may be considered pathological.
Change in upper limb function measured with QuickDASH questionnaire (score 0-100) | Baseline (before intervention), Immediately post-program (Day 0 after completion)
  Upper limb function will be measured with the DASH (Disabilities of the Arm, Shoulder, and Hand) questionnaire. This tool assesses the function of the arm, shoulder, and hand in patients with disorders or injuries in these areas. Responses are scored on a scale from 0 to 4, where 0 means no difficulty or pain, and 4 indicates severe difficulty or unbearable pain. The total score is calculated by summing responses and normalizing to a 0-100 scale, where 0 indicates no disability (perfect function) and 100 indicates maximum disability or total loss of function.
Change in range of motion of shoulder rotations, elbow and wrist flexion-extension measured with goniometer (degrees) | Baseline (before intervention), Immediately post-program (Day 0 after completion)
  Range of motion (shoulder rotations, elbow and wrist flexion-extension) will be measured using a manual goniometer, a clinical, physiotherapeutic, and biomechanical tool used to assess joint angles. Shoulder rotation movements will be evaluated, as well as flexion and extension for the elbow and wrist.
Change in quality of life from baseline measured with EORTC QLQ-C30 questionnaire (score 0-100) | Baseline (before intervention), Immediately post-program (Day 0 after completion)
  Quality of life will be assessed with the EORTC Breast Cancer-Specific Questionnaire (QLQ-BR23), a specific version of the EORTC QLQ-C30 designed to evaluate quality of life in women diagnosed with breast cancer. This questionnaire complements the EORTC QLQ-C30 by adding questions focused on symptoms and concerns specific to breast cancer patients, as well as side effects related to treatments. Each item is scored on a scale from 0 to 4, where a higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Aïda Cadellans Arróniz (Principal Investigator), PT, PhD, Principal Investigator — Universitat Internacional de Catalunya

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data (IPD) will be made available to qualified researchers upon reasonable request, following publication of the primary results. Data will be shared via institutional repository or secure data-sharing platform.
Supporting Information: Study Protocol
Time Frame: IPD will be shared at the time of publication of the main results and will be available for up to 5 years.
Access Criteria: Data will be shared with qualified researchers upon reasonable request for scientific purposes, subject to approval by the study team. A data access agreement will be required.
URL: https://zenodo.org/